CLINICAL TRIAL: NCT04784611
Title: Our Peers - Empowerment and Navigational Support: - A Peer Health Navigator Intervention for Medicaid Beneficiaries With Physical Disabilities
Brief Title: Our Peers - Empowerment and Navigational Support
Acronym: OP-ENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Shirley Ryan AbilityLab (Other); Oakland University (Other); Access Living (Unknown)
Responsible Party: Principal Investigator, Susan Magasi, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-1207
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Disabled Persons
Keywords: peer health navigator; community health worker

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention or usual care groups using block randomization with randomly selected blocks of 4, 8 or 12. Randomization sequence will be generated using SAS algorithm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the nature of the intervention it is not possible to mask participants and interventionists to group assignment. Outcome assessors and investigators will be unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - OP-ENS Intervention (Experimental): Participants will be matched with a peer health navigator. As part of this complex behavioral intervention, participants and peer health navigators will engage in a systematic process of barrier and strength identification, goal setting and action planning related to issues of healthcare access and quality. Participants and peers will meet at least monthly over the course of the 12-month study period (but frequency is determined by participant need). Given the nature of the disability and healthcare experience, we anticipate the needs and therefore frequency will fluctuate over the duration of the study period. Beginning in month 10, participants and peers will engage in a period of transition planning to ensure that participants have the strategies and supports in place to assume the role of their own health navigator.
  Interventions: Behavioral: Our Peers - Empowerment and Navigational Support (OP-ENS) Peer Health Navigator Intervention
- Group 2 - Usual Care (No Intervention): Participants randomized to the usual care group will continue with their usual health and healthcare routines. Participants in the usual care group will receive a monthly newsletter with general interest information relevant to the disability community.

INTERVENTIONS:
Behavioral: Our Peers - Empowerment and Navigational Support (OP-ENS) Peer Health Navigator Intervention — Disability peer health navigator mentored and manualized process of barriers identification, asset mapping, goal setting, and action planning along with on-going social support and information sharing.
  Arms: Group 1 - OP-ENS Intervention

SUMMARY:
People with physical disabilities experience well documented barriers to healthcare access, quality and outcomes. The purpose of this study is to implement and evaluate a 12-month peer health navigator intervention (called Our Peer-Empowerment and Navigational Support) designed to help Medicaid beneficiaries with physical disabilities break down barriers to care through a systematic process of 1) rapport building, 2) identification of healthcare needs and priorities, 3) identification of barriers and supports, 4) co-creation of goal and action plans, and 5) provision of social and informational support. It is hypothesized that people in the interventional trial will experience: improved patient activation, increased social support, increased access to care, increased quality of care, and increased health outcomes compared to people in the control group.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the preliminary effectiveness and social validity of the OP-ENS (Our Peers - Empowerment and Navigational Support). a 12-month peer health navigator intervention sing a clinical trial design in a sample of community-dwelling adult Medicaid beneficiaries with physical disabilities.

Participants will be recruited through community and clinical networks and screened for eligibility. Participants will be randomly assigned to either the intervention or usual care groups. Participants in the intervention group will be matched with a trained peer health navigator (who is also a person with a physical disability). Using a structure process of barrier identification, goal setting and action planning peer health navigators will work with participants to help address their healthcare needs and concerns, including such things as patient-provider communication, transportation, access to durable medical equipment. It is important to note that peer health navigators are not healthcare providers and do not provide medical or health advice. Participants in the intervention trial are asked to meet with their peer health navigator at least once a month during the study period. To encourage participation in this intervention, progressive micro-incentives are integrated into the study protocol. To promote equipoise, a similar micro-incentive schedule is created for the usual care group.

Data Collection - All participants, regardless of group assignment, will be interviewed at 3 time points (baseline, 6 months, 13 months) using a self-report measures of healthcare access, quality, and outcomes as well as measures of social support and patient activation. Data collectors will be blinded to group assignment and not involved in the delivery of the OP-ENS intervention.

Data Analysis - The investigators will employ mixed effects model using each study outcome as a time-varying dependent variable and treatment group (PHN vs. usual care) as the main fixed effect. Baseline characteristics including race/ethnicity, gender, and socioeconomic status will be entered as time-invariant covariates if baseline group differences are observed (in spite of randomization). Subject intercept will be modeled as a random effect. The null hypothesis will be rejected if a significant group*time interaction effect is observed. The investigators hypothesize that PHN will have a more favorable trajectory slope of study outcomes than the matched control group. For each hypothesis, post-hoc analysis will be conducted to assess difference in each outcome variable between the two groups at different time points. The mixed models will run using PROC MIXED from of SAS 9.3 (Cary, NC). The method of estimation will be maximum likelihood (ML). A variety of covariance structures (first order regressive, compound symmetry, toeplitz, variance components, unstructured) will be carefully examined and compared for best model fit, Akaike's Information (AIC) and Bayesian Information Criteria (BIC). These statistics are functions of the log likelihood and can be compared across models. As missing data are inevitable in a longitudinal study, values will be imputed where possible using either mean (median) substitute or formal imputation procedures such as EM algorithm if missing data are MCAR (missing completely at random) or MAR (missing at random). If missing data are NMAR (not missing at random), the "pattern mixture" approach will be used to compute a "weighted average" of the parameters that are associated with the missing data to estimate what the data would have been.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid beneficiary
* self-identified as person with a disability
* ability to provide legal consent
* ability to communicate in English

Exclusion Criteria:

* diagnosis of several persistent mental illness, substance abuse, primary diagnosis of pain with narcotic management.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Activation Measure (PAM) scores | baseline to 6-months
  13-item self-report measure of perceived knowledge, skills &confidence in self-management
Change in Health care access and quality using CAHPS - Adult Medicaid Survey 5.0 | baseline to 6-months
  Self-report measure of consumer's experiences, Composite scores - access and availability of care, experience of care, special considerations for people with disabilities.
Change in Patient Activation Measure (PAM) scores | baseline to 13-months
  13-item self-report measure of perceived knowledge, skills &confidence in self-management
Change in Health care access and quality using CAHPS - Adult Medicaid Survey 5.0 | baseline to 13-months
  Self-report measure of consumer's experiences, Composite scores - access and availability of care, experience of care, special considerations for people with disabilities.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Score | baseline to 6-months
  8-item self-report measure of an individual's physical, mental, and social health. Items are rated on a Likert-scale. The PROMIS Global scale produces a physical and a mental health score from 4 items each. (minimum raw score 4; maximum raw score 20 for each physical health and mental health.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score | baseline to 6-months
  8-item self-report measure of the consequences of pain on relevant aspects of life. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of pain interference.
Change in Patient Reported Outcomes Measurement Information Systems (PROMIS) Depression Score | baseline to 6-months
  8-item self-report measure of negative mood, views of self, and social cognition as well as decreased positive affect and engagement. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of emotional distress.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) fatigue | baseline to 6-months
  8-item self-report measure of the consequences of the experience and consequences of fatigue physical, mental and social activities. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of fatigue and fatigue impact.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Informational Support Score | baseline to 6-months
  8-item short form of perceived availability of helpful information or advice. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher availability of information support..
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Support Scores | baseline to 6-months
  8-item self report of perceived perceived feelings of being cared for and valued as a person. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of emotional support.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities Scores | baseline to 6-months
  8-item self-report of perceived ability to perform one's usual social roles and activities. 8-item self-report measure of the consequences of pain on relevant aspects of life. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of better ability to participate in social activities and roles.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Score | baseline to 13-months
  8-item self-report measure of an individual's physical, mental, and social health. Items are rated on a Likert-scale. The PROMIS Global scale produces a physical and a mental health score from 4 items each. (minimum raw score 4; maximum raw score 20 for each physical health and mental health.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score | baseline to 13-months
  8-item self-report measure of the consequences of pain on relevant aspects of life. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of pain interference.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) fatigue | baseline to 13-months
  8-item self-report measure of the consequences of the experience and consequences of fatigue physical, mental and social activities. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of fatigue and fatigue impact.
Change in Patient Reported Outcomes Measurement Information Systems (PROMIS) Depression Score | baseline to 13-months
  8-item self-report measure of negative mood, views of self, and social cognition as well as decreased positive affect and engagement. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of emotional distress.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Informational Support Score | baseline to 13-months
  8-item short form of perceived availability of helpful information or advice. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher availability of information support..
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Support Scores | baseline to 13-months
  8-item self report of perceived perceived feelings of being cared for and valued as a person. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of higher level of emotional support.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities Scores | baseline to 13-months
  8-item self-report of perceived ability to perform one's usual social roles and activities. 8-item self-report measure of the consequences of pain on relevant aspects of life. Each item is rated on a 5-point Likert scale. Minimum raw score = 8; maximum raw score = 40. Higher scores are indicative of better ability to participate in social activities and roles.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Magasi, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Chicago, Illinois, United States